CLINICAL TRIAL: NCT07059741
Title: A Prospective Study of Integrated Radiotherapy-optimized ASCT Sequential CAR-T Therapy on the Efficacy and Safety of Patients With Relapsed and Refractory Aggressive B-cell Non-Hodgkin Lymphoma.
Brief Title: Integrated Radiotherapy-optimized ASCT Sequential CAR-T Therapy for Patients With Relapsed and Refractory B-NHL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2024415
Record Dates: First submitted 2024-11-07; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Aggressive B-Cell Non-Hodgkin's Lymphoma (NHL)
Keywords: Radiotherapy; autologous stem cell transplantation; Relapsed and refractory; circulating tumor DNA; Chimeric antigen receptor T-cell therapy
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (PET/CT-, ctDNA+) (Experimental): Patients will receive low-dose radiotherapy (RT) combined with reduced-intensity SEAM/TB chemotherapy as a conditioning regimen, followed by autologous stem cell transplantation (ASCT) and sequential CAR-T cell therapy.
  Interventions: Other: integrated low-dose RT with reduced SEAM/TB conditioning before ASCT sequential CAR-T
- Cohort 2 (PET/CT+, ctDNA+) (Experimental): Patients will receive high-dose RT combined with reduced-intensity SEAM/TB chemotherapy as a conditioning regimen, followed by ASCT and sequential CAR-T cell therapy.
  Interventions: Other: integrated high-dose RT with reduced SEAM/TB conditioning before ASCT sequential CAR-T

INTERVENTIONS:
Other: integrated low-dose RT with reduced SEAM/TB conditioning before ASCT sequential CAR-T — 1. RT regimen:
     localized low dose RT: 1-1.5Gy/fraction*5fractions
  2. Reduced dose SEAM regimen (CNS uninvolved):
     * Simustine 250mg/m2 d-6 orally
     * Cytarabine 200mg/m2 q12h d-5~d-4 intravenous infusion
     * Etoposide 100mg/m2 q12h d-5~d-4 intravenous infusion
     * Melphalan 140mg/m2 q12h d-3 intravenous infusion
  3. TB regimen (CNS involvement):
     * Thiotepa 250mg/m2 qd, d-8~d-6 intravenous infusion
     * Busulfan 0.8mg/kg q6h d-5~d-3 intravenous infusion
  Arms: Cohort 1 (PET/CT-, ctDNA+)
Other: integrated high-dose RT with reduced SEAM/TB conditioning before ASCT sequential CAR-T — 1. RT regimen:
     localized high dose RT: 3-6Gy/fraction*5fractions
  2. Reduced dose SEAM regimen (CNS uninvolved):
     * Simustine 250mg/m2 d-6 orally
     * Cytarabine 200mg/m2 q12h d-5~d-4 intravenous infusion
     * Etoposide 100mg/m2 q12h d-5~d-4 intravenous infusion
     * Melphalan 140mg/m2 q12h d-3 intravenous infusion
  3. TB regimen (CNS involvement):
     * Thiotepa 250mg/m2 qd, d-8~d-6 intravenous infusion
     * Busulfan 0.8mg/kg q6h d-5~d-3 intravenous infusion
  Arms: Cohort 2 (PET/CT+, ctDNA+)

SUMMARY:
This study aims to investigate a novel therapeutic strategy of integrated radiotherapy before autologous stem cell transplantation (ASCT) sequential chimeric antigen receptor T-cell(CAR-T) therapy for patients with relapsed/refractory(R/R) aggressive B-cell non-Hodgkin lymphoma (B-NHL). By evaluating the efficacy and safety of this multimodal approach, we seek to provide a theoretical foundation and clinical data to optimize outcomes for relapsed/refractory aggressive B-NHL patients.

DETAILED DESCRIPTION:
This trial will enroll R/R aggressive B-NHL patients aged ≥18 years who have undergone at least two prior lines of systemic therapy. Participants will be stratified into two cohorts based on post-salvage therapy disease status:

Cohort 1 (PET/CT-, ctDNA+): Patients will receive low-dose radiotherapy (RT) combined with reduced-intensity SEAM/TB chemotherapy as a conditioning regimen, followed by ASCT and sequential CAR-T therapy.

Cohort 2 (PET/CT+, ctDNA+): Patients will receive high-dose RT combined with reduced-intensity SEAM/TB chemotherapy as a conditioning regimen, followed by ASCT and sequential CAR-T therapy.

All patients completing the combined ASCT-CAR-T protocol will undergo longitudinal follow-up for safety, efficacy survival outcomes .

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Histologically confirmed aggressive B-NHL.
3. Life expectancy >3 months.
4. Appropriate organ function:

   Cardiac function: cardiac ejection fraction ≥50%; Liver function: alanine aminotransferase and glutamic aminotransferase ≤ 2 times the upper limit of normal values; renal function: serum creatinine clearance ≥80 mL/min; serum creatinine <160 mmol/L Lung function: SPO2>91% without oxygen intake
5. Adequate bone marrow reserve defined as:

   hemoglobin ≥90 g/L. platelet count ≥70 x 10^9/L. absolute neutrophil count ≥1.5 x 10^9/L.
6. The patient is capable of understanding and willing to provide written informed consent.
7. Subjects of childbearing or childbearing potential must be willing to practice birth control from the date of enrollment in this study until study follow-up.

Exclusion Criteria:

1. severe hepatic and renal function abnormalities (alanine aminotransferase, bilirubin, creatinine > 2 times the upper limit of normal);
2. Presence of organic heart disease with resulting clinical symptoms or abnormal cardiac function (NYHA cardiac function classification ≥ grade 2);
3. ECG QTc interval >500 ms;
4. active hepatitis B/hepatitis C;
5. uncontrolled active infection;
6. human immunodeficiency virus infection;
7. concurrent other tumors requiring treatment or intervention;
8. current or anticipated need for systemic corticosteroid therapy;
9. pregnant or lactating women;
10. abandonment of consolidation autologous hematopoietic stem cell transplantation for financial reasons;
11. other psychological conditions that prevent the patient from participating in the study or signing the informed consent form;
12. Subjects who, in the judgment of the investigator, are unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or do not meet the requirements for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2028-12-10 (Estimated); Study Completion 2028-12-10 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate(CRR) | At the end of 3 months after CAR-T infusion
  The rate of patients who achieved CR 3 months after CAR-T infusion

SECONDARY OUTCOMES:
Major adverse reactions | From enrollment to 1 month after CAR-T infusion of last patient
  The safety and tolerability of the therapeutic regimen measured by the major adverse events.
Time to bone marrow hematopoietic reconstitution | From enrollment to 3 months after stem cell infusion of last patient
  The time of bone marrow hematopoietic reconstitution after stem cell infusion
2-year progression-free survival(PFS) | From enrollment to 2-year after the end of last patient's treatment
  PFS will be assessed from the first date of radiotherapy to the progression of the disease, death, or last follow-up.
2-year overall survival(OS) | From enrollment to 2-year after the end of last patient's treatment
  OS will be assessed from the first date of radiotherapy to death from any cause or last follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No